CLINICAL TRIAL: NCT01373190
Title: Thermographic Examination of Low Back and Abdominal Area Skin Temperatures in Individuals With and Without Focal Onset Epilepsy
Brief Title: Thermographic Examination of Skin Temperatures in Individuals With Focal Onset Epilepsy
Status: Completed | Type: Observational
Sponsor: Atlantic University (Other)
Collaborators: A.T. Still University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hollis King, Professor, University of Wisconsin, Madison
Other Study IDs: AU Epilepsy Study
Record Dates: First submitted 2011-06-02; First posted 2011-06-14 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Focal Onset Epilepsy; Partial Epilepsy
Keywords: epilepsy; thermography
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epilepsy Group: Individuals diagnosed with Partial/Focal Onset Epilepsy ICD9CM 345.4 and/or 345.5
- Control Group: Individuals who do not have the diagnosis of Epilepsy and have no history of seizure disorders

SUMMARY:
The specific aim is to determine if there are patterns of temperature differences in the abdominal and back regions of individuals with partial/focal onset epilepsy as compared to a non-epileptic control group. The hypothesis is that individuals with partial/focal onset epilepsy will have colder recorded temperatures in the abdominal area than individuals in a matched control group.

DETAILED DESCRIPTION:
The concept of "Abdominal Epilepsy" has been described in the neurology literature. The present study seeks to amplify understanding of this clinical entity by measuring abdominal area and low back skin temperature changes which may be affected through the function of the abdominal ganglia, specifically the Celiac, Superior Mesenteric and Inferior Mesenteric Ganglia.

This not an intervention study. It is study comparing abdominal area and low back skin temperature in individuals with the Partial/Focal Onset Epilepsy with a match control group of individuals with no epilepsy history. The implications of the outcome of the finding any significant temperature changes between the experimental and control groups is great enough to warrant the highest level of scientific scrutiny that this registration permits.

ELIGIBILITY:
Inclusion Criteria Experimental Group:

1. Diagnosis of Partial/Focal Onset Epilepsy (ICD9-CM 345.4 and 345.5)
2. Ages 18-70

Exclusion Criteria Experimental Group:

1. Pregnancy
2. Recent trauma such as motor vehicle accident or injury to the musculoskeletal system
3. Currently on medication, other than for epilepsy which may affect autonomic nervous system function, e.g. Glaucoma medication
4. If diagnosed with a condition which could affect abdominal area neurophysiologic functions.

   1. Irritable bowel syndrome
   2. Crohn's disease
   3. Ulcerative colitis
   4. Migraine headache with abdominal manifestation

Inclusion criteria Control group:

1. No history or diagnosis of any seizure disorder
2. Ages 18-70

Exclusion Criteria Control group:

1. Pregnancy
2. Recent trauma such as motor vehicle accident or injury to the musculoskeletal system
3. Currently on medication, other than for epilepsy which may affect autonomic nervous system function, e.g. Glaucoma medication
4. If diagnosed with a condition which could affect abdominal area neurophysiologic functions.

   1. Irritable bowel syndrome
   2. Crohn's disease
   3. Ulcerative colitis
   4. Migraine headache with abdominal manifestation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 individual with diagnosis of focal onset epilepsy 50 normal matched control subjects
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Thermographic imagery of the abdominal area | Each experimental subject and each control subject will be seen once for the administration of the thermography imagery
  State of the art thermographic imagery of the imagery of the abdominal area from the xyphoid bone to just above the public symphysis. It is hypothesized that the average temperature for the experimental group will be lower than the control group. Since this is a measurement or diagnostic study using thermographic imagery, there is no health risk to the subjects.

SECONDARY OUTCOMES:
low back thermography imagery | one time for thermographic imagery
  Besides abdominal area will also do theographic imagery of low back of subjects because of the possibility of dermatomal skin area temperature changes possibly related the "Abdominal Epilepsy" dysfunction of the Celiac, Superior Mesenteric and Inferior Mesenteric Ganglia
side thermography imagery | one time for thermographic imagery
  To capture possible dermatomal skin temperature effects will do thermographic imagery of the side or lateral aspect of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Hollis H King, DO, PhD, Principal Investigator — AT Still University of Health Sciences
Locations (1):
- Epilepsy Foundation of Florida, Miami, Florida, United States

REFERENCES:
- [Background] Henkel A, Noachtar S, Pfander M, Luders HO. The localizing value of the abdominal aura and its evolution: a study in focal epilepsies. Neurology. 2002 Jan 22;58(2):271-6. doi: 10.1212/wnl.58.2.271. PMID 11805256
- [Background] Zinkin NT, Peppercorn MA. Abdominal epilepsy. Best Pract Res Clin Gastroenterol. 2005 Apr;19(2):263-74. doi: 10.1016/j.bpg.2004.10.001. PMID 15833692